CLINICAL TRIAL: NCT03205137
Title: Comparison of the Medication Adherence of Patients Treated With Telmisartan/Hydrochlorothiazide or Telmisartan/Amlodipine Fixed Dose Combination (FDC) Versus Double-pill Combination Therapy Based on Database Data in Real-world Japanese Therapeutic Practice
Brief Title: Comparison of the Medication Adherence of Patients Treated With Telmisartan/Hydrochlorothiazide or Telmisartan/Amlodipine Fixed Dose Combination (FDC) Versus Double-pill Combination Therapy in Real-world Japanese Therapeutic Practice
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0502-0612
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Telmisartan and hydrochlorothiazide group
  Interventions: Drug: subjects treated with telmisartan/hydrochlorothiazide
- Telmisartan and amlodipine group
  Interventions: Drug: Subjects treated with Telmisartan and amlodipine
- Telmisartan+hydrochlorothiazide double-pill combination group
  Interventions: Drug: subjects treated with Telmisartan+hydrochlorothiazide double-pill combination group
- telmisartan+amlodipine double-pill combination group
  Interventions: Drug: subjects treated with telmisartan+amlodipine double pill

INTERVENTIONS:
Drug: subjects treated with telmisartan/hydrochlorothiazide — subjects treated with telmisartan/hydrochlorothiazide
  Other Names: MICARDIS, PRITOR, TELMISARTAN
  Groups: Telmisartan and hydrochlorothiazide group
Drug: Subjects treated with Telmisartan and amlodipine — Subjects treated with Telmisartan and amlodipine
  Other Names: MICARDIS, PRITOR, TELMISARTAN
  Groups: Telmisartan and amlodipine group
Drug: subjects treated with Telmisartan+hydrochlorothiazide double-pill combination group — subjects treated with Telmisartan+hydrochlorothiazide double-pill combination group
  Other Names: MICARDIS, PRITOR, TELMISARTAN
  Groups: Telmisartan+hydrochlorothiazide double-pill combination group
Drug: subjects treated with telmisartan+amlodipine double pill — subjects treated with telmisartan+amlodipine double pill
  Other Names: MICARDIS, PRITOR, TELMISARTAN
  Groups: telmisartan+amlodipine double-pill combination group

SUMMARY:
The primary objective of this study is to compare the medication adherence measured by PDC of patients with FDC or double-pill combination therapy in real-world Japanese therapeutic practice.The further objective of this study is how much influence the background of patients to the adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension
* Patients must have their first prescription (defined as index date*) for telmisartan and hydrochlorothiazide or Micombi® between 01/07/2010 and 28/09/2010
* Patients must have their first prescription (defined as index date*) for telmisartan and amlodipine or Micamlo® between 10/12/2010 and 09/03/2011
* Patients must have at least 180 days follow up verified by the presence of prescription record

Exclusion Criteria:

* Patients who were under 40 years old at the time of enrolment
* Patients who prescribed the study drugs less than 90 days during a follow up period of 180 days
* Patients whose visits are less than 2 times during a follow up period of 180 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Japan Medical Information Research Institute (JMIRI), Inc. prescription database is used.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-07-11 (Estimated); Study Completion 2022-07-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of days covered of patients treated with single- and double- combination therapy | 180 days

SECONDARY OUTCOMES:
Demographic and clinical characteristics of patients treated with single- and double combination | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com